CLINICAL TRIAL: NCT01541917
Title: WebSMART: Efficacy of Web-based Pain Self-management for Adolescents With Juvenile Idiopathic Arthritis
Brief Title: Efficacy of Web-based Pain Self-management for Adolescents With Juvenile Idiopathic Arthritis
Acronym: WebSMART
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Children's Mercy Hospital Kansas City (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GRANT10829275; 1R01AR061513-01 (NIH)
Record Dates: First submitted 2012-02-24; First posted 2012-03-01 (Estimated); Results first posted 2017-03-09 (Actual); Last update posted 2017-03-09 (Actual); Status verified 2017-01

CONDITIONS: Juvenile Idiopathic Arthritis
MeSH Terms: conditions — Arthritis, Juvenile

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Web-based coping skills training (Experimental): Involves completion of a 12-week interactive, multi-component, multimedia online training that consists of instruction in specific self-management strategies, disease education, and social support.
  Interventions: Behavioral: Web-based coping skills training
- Online disease education (Active Comparator): Involves viewing 12 educational websites about Juvenile Idiopathic Arthritis over the course of 12 weeks.
  Interventions: Behavioral: Online disease education

INTERVENTIONS:
Behavioral: Web-based coping skills training — This intervention comprises a 12-week interactive, multi-component, multimedia online training that consists of instruction in specific self-management strategies, disease education, and social support. The content is rooted in cognitive-behavioral principles of disease self-management. In addition to the web-based modules, the intervention consists of monthly telephone support for 3 months by a trained bilingual health coach (research nurse) to review material and help enhance motivation.
  Arms: Web-based coping skills training
Behavioral: Online disease education — The online disease education intervention provides access to an online resource center containing links to 12 educational websites about Juvenile Idiopathic Arthritis. Participants will be asked to review one educational website per week over the course of 12 weeks. Participants also will receive three monthly phone calls by a bilingual nurse "health coach" to discuss the participant's efforts at managing his/her disease.
  Arms: Online disease education

SUMMARY:
The purpose of this multi-site randomized clinical trial is to determine if an online coping skills training program will produce superior improvements in pain and health-related quality of life outcomes for adolescents with JIA relative to outcomes attained with reviewing online educational information about JIA.

DETAILED DESCRIPTION:
There is a critical gap in the contemporary treatment of Juvenile Idiopathic Arthritis (JIA) wherein a majority of adolescent patients still experience ongoing pain and reduced health-related quality of life even with advances in medical management of the disease. Despite the pervasiveness of this problem, most adolescents receive no training in the strategies that can help empower them to reduce pain and disability. The Internet offers a unique opportunity to reach adolescents with JIA and provide the training in pain self-management strategies that otherwise may not occur due to treatment access and resource obstacles. The objective of this research study is to conduct a definitive test of an investigator-developed online coping skills training program for English- and Spanish-speaking adolescents with JIA. Based on data from the investigators' preliminary work, the central hypothesis is that use of an online coping skills training program will produce superior improvements in pain and health-related quality of life outcomes for adolescents with JIA relative to outcomes attained with reviewing extant online educational information about JIA and receiving additional attention to coping efforts (control condition). Specific aims for the proposed work include (a) determining the extent to which an online coping skills training program for adolescents with JIA produces improvements in key health outcomes that currently do not optimally respond to only contemporary medical management (pain and health-related quality of life); and (b) determining predictors of change in pain and health-related quality of life indices in adolescents with JIA and establishing the extent to which online coping skills training influences health outcomes via these predictors. An exploratory aim is to determine the acceptability and preliminary efficacy of online coping skills training within a subgroup of Hispanic adolescents with JIA. These aims will be achieved through the approach of using a multi-center randomized controlled trial in which a sample of 360 consenting English- and Spanish-speaking adolescents aged 12-18 years with JIA will be enrolled and randomized into one of two groups: (a) an experimental group consisting of a 12-week interactive online multi-component treatment protocol including targeted disease education, training in empirically supported cognitive-behavioral coping skills, and social support augmented by monthly telephone contact with a nurse; or (b) a control group consisting of 12 weeks of guided access to extant online resources for disease education and additional attention to own best efforts at managing JIA via monthly telephone contact with a nurse. Outcome data will be collected from both groups prior to treatment, immediately following the intervention, and at 6- and 12-month follow-up assessments. Successful completion of this project is expected to establish to what extent and how an innovative online self-management program produces change in clinically relevant health outcomes in both English- and Spanish-speaking adolescents with JIA. The proposed study therefore can be expected to have a significant positive impact in the healthcare of teens with JIA and in identifying treatment targets for other youth self-management interventions.

ELIGIBILITY:
Inclusion Criteria:

* 12-18 years of age (inclusive)
* diagnosed with JIA by a pediatric rheumatologist
* able to speak and read English and/or Spanish
* able to complete online measures
* reporting pain in at least one joint over the past 6 months

Exclusion Criteria:

* have another chronic medical condition that adversely impacts pain and/or health-related quality of life (e.g., inflammatory bowel disease, fibromyalgia, cancer, genetic disorder, pervasive developmental disorder, diabetes)
* have a significant cognitive impairment or illiteracy that would prevent understanding of the intervention and outcome measures
* currently in psychotherapy

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 305 (Actual)
Dates: Start 2012-07; Primary Completion 2016-04 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark A Connelly, PhD, Principal Investigator — Children's Mercy Hospital Kansas City; Jennifer Stinson, PhD, Principal Investigator — The Hospital for Sick Children
Locations (10):
- United States (10):
  - University of California San Francisco Benioff Children's Hospital, San Francisco, California
  - Lurie Children's Hospital, Chicago, Illinois
  - Riley Hospital for Children, Indianopolis, Indiana
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Joseph M. Sanzari Children's Hospital, Hackensack, New Jersey
  - Duke University Medical Center, Durham, North Carolina
  - Nationwide Children's Hospital, Columbus, Ohio
  - The Children's Hospital at Legacy Emmanuel Medical Center, Portland, Oregon
  - Dell Children's Medical Center of Central Texas, Austin, Texas
  - Seattle Children's Hospital, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
A deidentified dataset is available for secondary analyses per our Resource Sharing Plan.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: For this trial, 305 patients consented (were enrolled) to participate, but 7 of these patients subsequently were found to not fully meet eligibility criteria and 9 of these patients dropped out prior to being randomized. The total randomized sample therefore is 289.
Groups:
- Online Disease Education Control: Involves viewing 12 educational websites about Juvenile Idiopathic Arthritis over the course of 12 weeks.
  Online disease education: The online disease education intervention provides access to an online resource center containing links to 12 educational websites about Juvenile Idiopathic Arthritis. Participants will be asked to review one educational website per week over the course of 12 weeks. Participants also will receive three monthly phone calls by a bilingual nurse "health coach" to discuss the participant's efforts at managing his/her disease.
Period: Overall Study
Arm/Group | Web-based Coping Skills Training | Online Disease Education Control
Started | 144 | 145
Completed | 129 | 136
Not Completed | 15 | 9
Not completed — Lost to Follow-up | 2 | 2
Not completed — Withdrawal by Subject | 13 | 7

BASELINE CHARACTERISTICS:
Groups:
- Web-based Coping Skills Training: This intervention comprises a 12-week interactive, multi-component, multimedia online training that consists of instruction in specific self-management strategies, disease education, and social support. The content is rooted in cognitive-behavioral principles of disease self-management. In addition to the web-based modules, the intervention consists of monthly telephone support for 3 months by a trained bilingual health coach to review material and help enhance motivation.
- Online Disease Education Control: The online disease education intervention provides access to an online resource center containing links to 12 educational websites about Juvenile Idiopathic Arthritis. Participants will be asked to review one educational website per week over the course of 12 weeks. Participants also will receive three monthly phone calls by a bilingual health coach to discuss the participant's efforts at managing his/her disease.
- Never Randomized: This group comprises participants that consented but were never randomized to a condition due to being determined to not meet eligibility criteria or self-withdrawing before randomization.
- Total: Total of all reporting groups
Arm/Group | Web-based Coping Skills Training | Online Disease Education Control | Never Randomized | Total
Number analyzed (Participants) | 144 | 145 | 16 | 305
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.65 (1.85) | 14.55 (1.76) | 15.06 (1.69) | 14.59 (1.79)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 98 | 111 | 13 | 222
  Male | 46 | 34 | 3 | 83
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 21 | 17 | 1 | 39
  Not Hispanic or Latino | 123 | 128 | 15 | 266
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 0 | 0 | 3
  Asian | 5 | 5 | 0 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 2 | 0 | 2
  Black or African American | 7 | 5 | 1 | 13
  White | 120 | 123 | 13 | 256
  More than one race | 9 | 10 | 2 | 21
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Pain Intensity
Description: Pain intensity was assessed by patient-self report using an electronic numeric rating scale ranging from 0-10, with 0 being the lowest value ("no pain") and 10 being the highest value ("very much pain").
Time Frame: Baseline, post-treatment, 6-month follow-up, 12-month follow-up
Population: All randomized patients were analyzed regardless of whether or not they completed treatment (intent to treat analyses).
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- Online Disease Education Control: The online disease education intervention provides access to an online resource center containing links to 12 educational websites about Juvenile Idiopathic Arthritis. Participants will be asked to review one educational website per week over the course of 12 weeks. Participants also will receive three monthly phone calls by a bilingual nurse "health coach" to discuss the participant's efforts at managing his/her disease.
Arm/Group | Web-based Coping Skills Training | Online Disease Education Control
Number analyzed (Participants) | 144 | 145
Units on a scale
  Baseline | 3.56 (2.33) | 3.26 (2.38)
  Post-Treatment | 3.07 (2.47) | 2.90 (2.45)
  6-Month Follow-Up | 2.87 (2.45) | 2.96 (2.29)
  12-Month Follow-Up | 3.07 (2.49) | 2.71 (2.43)
Statistical Analysis 1: Comparison: Web-based Coping Skills Training vs Online Disease Education Control; Multilevel growth model evaluating average change over time (regardless of group) on the outcome variable; Test type: Superiority or Other; p < .001, Multilevel growth model; Adjusted for baseline values; Slope = -.04, 95% CI 2-sided [-.06 to -.02], Standard Error of Mean .01 — The parameter represents the average monthly change on the outcome variable since group procedures were initiated
Statistical Analysis 2: Comparison: Web-based Coping Skills Training vs Online Disease Education Control; Multilevel linear growth modeling was used for analyses, with the time variable coded as months since randomization. All models included an adjustment for baseline group differences on the outcome variable; Test type: Superiority or Other; p = .51, Multilevel growth model; Slope = -.014, 95% CI 2-sided [-.055 to .027], Standard Error of Mean .021 — The estimated parameter value represents the difference in the monthly change (since baseline) in the outcome variable attributed to being in the treatment group (web-based coping skills training) versus the control group (online disease education)

2. Primary Outcome: Change in PedsQL Rheumatology Health-Related Quality of Life Total Score
Description: Health-related quality of life was measured by patient self-report using an electronic version of the PedsQL Rheumatology Module. Responses on this scale are transformed into a 0-100 scale, with 0 being the worst value for health-related quality of life and 100 being the best possible value for health-related quality of life.
Time Frame: Pre-intervention, post-intervention, 6-month follow-up, 12-month follow-up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Web-based Coping Skills Training | Online Disease Education
Number analyzed (Participants) | 144 | 145
units on a scale
  Baseline | 72.56 (15.52) | 72.44 (15.81)
  Post-Treatment | 75.68 (16.68) | 77.78 (15.02)
  6-Month Follow-Up | 77.32 (15.64) | 77.12 (14.41)
  12-Month Follow-Up | 78.26 (16.23) | 78.04 (14.33)
Statistical Analysis 1: Comparison: Web-based Coping Skills Training vs Online Disease Education; Multilevel growth model evaluating average change over time on the outcome variable; Test type: Superiority or Other; p < .001, Multilevel growth model; Adjusted for baseline values; Slope = .37, 95% CI 2-sided [.27 to .46], Standard Error of Mean .05 — The parameter represents the average monthly change on the outcome variable since before group procedures were started
Statistical Analysis 2: Comparison: Web-based Coping Skills Training vs Online Disease Education; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = .59, Multilevel growth model; Adjusted for baseline values on the outcome variable; Slope = .053, 95% CI 2-sided [-.144 to .252], Standard Error of Mean .101 — [estimate comment as in outcome 1, analysis 2]

3. Secondary Outcome: Change in Medical Issues, Exercise, Pain and Social Support Questionnaire (MEPS) Education Score
Description: Knowledge about Juvenile Idiopathic Arthritis was measured by patient self-report using an electronic version of the Medical Issues, Exercise, Pain and Social support (MEPS) Questionnaire. Responses on this scale are measured on a 0-10 numeric rating scale and averaged together to form a summary score, with 0 being the worst possible score and 10 being the best possible score.
Time Frame: Pre-intervention, post-intervention, 6-month follow-up, 12-month follow-up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Web-based Coping Skills Training | Online Disease Education
Number analyzed (Participants) | 144 | 145
units on a scale
  Baseline | 4.78 (2.35) | 4.57 (2.20)
  Post-Treatment | 6.27 (2.35) | 6.54 (2.03)
  6-Month Follow-Up | 6.62 (2.47) | 6.44 (2.40)
  12-Month Follow-Up | 6.45 (2.62) | 6.65 (2.28)
Statistical Analysis 1: Comparison: Web-based Coping Skills Training vs Online Disease Education; Multilevel growth model evaluating average change over time on the outcome variable; Test type: Superiority or Other; p < .001, Multilevel growth model; Adjusted for baseline values; Slope = .12, 95% CI 2-sided [.10 to .14], Standard Error of Mean .01 — The parameter represents the average monthly change on the outcome variable since before group procedures were started
Statistical Analysis 2: Comparison: Web-based Coping Skills Training vs Online Disease Education; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = .63, Multilevel growth model; Adjusted for baseline values on the outcome variable; Slope = -.01, 95% CI 2-sided [-.05 to .03], Standard Error of Mean .02 — [estimate comment as in outcome 1, analysis 2]

4. Secondary Outcome: Change in Disease Activity
Description: Disease activity was assessed by the treating physician based on a complete joint count (count of the number of joints that are swollen, painful, tender, or restriction in motion). The lowest (best) value is 0, and the highest (worst) possible value is 300.
Time Frame: Pre-intervention, post-intervention, 6-month follow-up, 12-month follow-up
Measure: Mean (Standard Deviation); unit: joints
Arm/Group | Web-based Coping Skills Training | Online Disease Education Control
Number analyzed (Participants) | 144 | 145
joints
  Baseline | 6.97 (12.84) | 6.63 (11.18)
  Post-Treatment | 5.61 (9.69) | 6.43 (10.09)
  6-Month Follow-Up | 5.45 (8.29) | 5.35 (8.14)
  12-Month Follow-Up | 4.53 (7.68) | 6.17 (9.90)
Statistical Analysis 1: Comparison: Web-based Coping Skills Training vs Online Disease Education Control; Multilevel growth model evaluating average change over time on the outcome variable; Test type: Superiority or Other; p = .02, Multilevel growth model; Adjusted for baseline values; Slope = -.10, 95% CI 2-sided [-.18 to -.01], Standard Error of Mean .04 — The parameter represents the average monthly change on the outcome variable since before group procedures were started
Statistical Analysis 2: Comparison: Web-based Coping Skills Training vs Online Disease Education Control; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = .91, Multilevel growth model; Adjusted for baseline values on the outcome variable; Slope = -.009, 95% CI 2-sided [-.174 to .155], Standard Error of Mean .084 — [estimate comment as in outcome 1, analysis 2]

5. Secondary Outcome: Change in Children's Arthritis Self-Efficacy (CASE) Scores
Description: Confidence in managing arthritis was measured by patient self-report using an electronic version of the Children's Arthritis Self-Efficacy (CASE) scale. Responses on a 5-point scale ("not at all sure" to "very sure") are averaged together to form a total score, with 0 being the worst possible value and 5 being the best possible value.
Time Frame: Pre-intervention, post-intervention, 6-month follow-up, 12-month follow-up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Web-based Coping Skills Training | Online Disease Education Control
Number analyzed (Participants) | 144 | 145
units on a scale
  Baseline | 3.31 (.96) | 3.32 (1.05)
  Post-Treatment | 3.80 (.88) | 3.67 (.99)
  6-Month Follow-Up | 3.81 (.94) | 3.73 (1.0)
  12-Month Follow-Up | 3.75 (.96) | 3.81 (.98)
Statistical Analysis 1: Comparison: Web-based Coping Skills Training vs Online Disease Education Control; Multilevel growth model evaluating average change over time on the outcome variable; Test type: Superiority or Other; p < .001, Multilevel growth model; Adjusted for baseline values; Slope = .0316, 95% CI 2-sided [.02 to .04], Standard Error of Mean .004 — The parameter represents the average monthly change on the outcome variable since before group procedures were started
Statistical Analysis 2: Comparison: Web-based Coping Skills Training vs Online Disease Education Control; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = .67, Multilevel growth model; Adjusted for baseline values on the outcome variable; Slope = -.004, 95% CI 2-sided [-.02 to .013], Standard Error of Mean .008 — [estimate comment as in outcome 1, analysis 2]

6. Secondary Outcome: Change in Approach Coping
Description: Scores on the Approach Coping sub-scale of the Pain Coping Questionnaire were used to measure approach coping, which is a type of coping considered to be adaptive and helpful for pain. Responses to items on this subscale are on a 5-point scale ("never use" to "very often use") and are averaged together for the subscale score, such that scores range from a worst possible value of 1 to a best possible value of 5.
Time Frame: Pre-intervention, post-intervention, 6-month follow-up, 12-month follow-up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Web-based Coping Skills Training | Online Disease Education Control
Number analyzed (Participants) | 144 | 145
units on a scale
  Baseline | 2.63 (.75) | 2.57 (.73)
  Post-Treatment | 2.84 (.87) | 2.67 (.88)
  6-Month Follow-Up | 2.76 (.90) | 2.55 (.87)
  12-Month Follow-Up | 2.71 (1.03) | 2.55 (.88)
Statistical Analysis 1: Comparison: Web-based Coping Skills Training vs Online Disease Education Control; Multilevel growth model evaluating average change over time on the outcome variable; Test type: Superiority or Other; p = .58, Multilevel growth model; Adjusted for baseline values; Slope = -.002, 95% CI 2-sided [-.01 to .01], Standard Error of Mean .004 — The parameter represents the average monthly change on the outcome variable since before group procedures were started
Statistical Analysis 2: Comparison: Web-based Coping Skills Training vs Online Disease Education Control; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = .49, Multilevel growth model; Adjusted for baseline values on the outcome variable; Slope = .005, 95% CI 2-sided [-.009 to .018], Standard Error of Mean .007 — [estimate comment as in outcome 1, analysis 2]

ADVERSE EVENTS:
Time Frame: Adverse events were monitored throughout participants' active participation in the trial, through 12 month follow-up.
Description: Information on adverse events were collected at each study visit (post-treatment, 6-month follow-up, 12-month follow-up) using a standardized electronic form.
Arm/Group | Web-based Coping Skills Training | Online Disease Education Control
Serious Adverse Events (participants affected / at risk) | 4/144 | 5/145
Other Adverse Events (participants affected / at risk) | 38/144 | 34/145
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Web-based Coping Skills Training (N=144) | Online Disease Education Control (N=145)
Hospitalization (Gastrointestinal disorders) | 1 (1) | 3 (4) — Hospitalized for evaluation of abdominal pain.
Arthritis flare (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Admitted to hospital for management of arthritis flare
Hospitalized for macrophage activation syndrome (Infections and infestations) | 0 (0) | 1 (1)
Hospitalized for appendicitis (Infections and infestations) | 0 (0) | 1 (1)
Hospitalized for management of Crohn's disease flare (Immune system disorders) | 1 (1) | 0 (0)
Hospitalized for suicidal thoughts (Psychiatric disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Web-based Coping Skills Training (N=144) | Online Disease Education Control (N=145)
Skin system findings (psoriasis, rash) (Skin and subcutaneous tissue disorders) | 5 (6) | 3 (4)
Injury (e.g., sprain, fracture) (Injury, poisoning and procedural complications) | 2 (2) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 7 (8)
Infection (Infections and infestations) | 7 (7) | 11 (11)
Blood disorder/problems (Blood and lymphatic system disorders) | 3 (3) | 2 (2)
Dizziness and/or fatigue (Nervous system disorders) | 2 (2) | 2 (2)
Arthritis flare (Immune system disorders) | 13 (18) | 4 (4)
Depression (Psychiatric disorders) | 3 (3) | 1 (1)
Suicidal thoughts (Psychiatric disorders) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No